CLINICAL TRIAL: NCT01949740
Title: Patient Preferences in Head and Neck Cancer Treatment Decisions - a Pilot Study of the Durability of Patient Priorities
Brief Title: Patient Preferences in Making Treatment Decisions in Patients With Stage I-IVA Oropharyngeal Cancer
Status: Terminated | Type: Observational
Why Stopped: Poor accrual
Sponsor: University of Chicago (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 13-0552; NCI-2013-01181 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); IRB13-0552; P30CA014599 (NIH)
Record Dates: First submitted 2013-09-20; First posted 2013-09-24 (Estimated); Last update posted 2015-09-02 (Estimated); Status verified 2015-09

CONDITIONS: Stage I Squamous Cell Carcinoma of the Oropharynx; Stage II Squamous Cell Carcinoma of the Oropharynx; Stage III Squamous Cell Carcinoma of the Oropharynx; Stage IVA Squamous Cell Carcinoma of the Oropharynx; Tongue Cancer
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Tongue Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Observational (patient preferences): Patients participate in a 45-minute interview comprising assessment of priorities and quality of life at baseline, 1, 6, and 12 months.
  Interventions: Other: questionnaire administration; Procedure: quality-of-life assessment

INTERVENTIONS:
Other: questionnaire administration — Ancillary studies
Procedure: quality-of-life assessment — Ancillary studies
  Other Names: quality of life assessment

SUMMARY:
This pilot research trial studies patient preferences in making treatment decisions in patients with stage I-IVA oropharyngeal cancer. Questionnaires that measure patient priorities before and after treatment may improve the ability to plan for better quality of life in patients with oropharyngeal cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the stability of Head and Neck Priorities Scale (HNPS) ranking between pre- and post-treatment assessments.

SECONDARY OBJECTIVES:

I. Use patient-interviews to refine and modify the HNPS for use in a larger scale trial.

II. Pilot the Head and Neck Patient Outcomes Survey (HNPOS) as a potential tool to identify priorities most important to quality-of-life outcomes.

III. Use the Functional Assessment of Cancer Therapy - Head and Neck (FACT-H&N) and EurolQoL-5D to determine the validity of the HNPOS.

OUTLINE:

Patients participate in a 45-minute interview comprising assessment of priorities and quality of life at baseline, 1, 6, and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Treatment naïve American Joint Committee on Cancer (AJCC) stage I-IVa squamous cell carcinoma of the head and neck with no definitive evidence of metastatic disease
* Sufficient vision, writing, and communication ability to complete the interviews and assessment tool
* Signed informed consent

Exclusion Criteria:

* Patients who are enrolled in other head and neck cancer treatment protocols are permitted to participate in this study if a) the other protocol permits this and b) the other protocol does not utilize the HNPS
* Patients who have previously undergone cancer treatment or are presently undergoing additional cancer treatments
* Patients who have already undergone unsuccessful curative-intent surgery on their head and neck cancer
* Patients, who have had a major surgery (defined as requiring general anesthesia but not including tonsillectomy, neck dissection, or panendoscopy [triple endoscopy or examination under general anesthesia]), or significant traumatic injury within 4 weeks of the study; patients who have not recovered from the side effects of any of the above surgeries
* Patients unwilling to or unable to comply with the protocol
* Patients unable to communicate with the interviewer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects will be identified through the Hematology/Oncology and ENT clinics a at their first visit for newly diagnosed Head/ Neck Cancer
Sampling Method: Non-Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2013-06; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Stability of HNPS ranking between pre- and post-treatment assessments | Up to 12 months
  Proportion of patients for whom the domain was considered stable calculated. Exact binomial tests will be used to test whether each proportion is greater than 50%.

SECONDARY OUTCOMES:
Reliability of HNPPQ scale, in terms of test-retest and internal consistency | Up to 12 months
  Weighted kappa coefficients will serve as the measure of agreement between the two replicates. Cronbach's alpha will be used to assess internal consistency.
Validity of HNPOS | Up to 12 months
  Nine HNPOS items will be compared to corresponding items on the FACT H&N scale. For each item, Kendall's tau-c will be computed for a measure of association suitable for contingency analyses of two ordinal variables.

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Langerman, Principal Investigator — University of Chicago Comprehensive Cancer Center
Locations (1):
- University of Chicago Comprehensive Cancer Center, Chicago, Illinois, United States